CLINICAL TRIAL: NCT03861000
Title: Evaluation of a Novel PET Radioligand for Phosphodiesterase-4D (PDE4D)
Brief Title: Title: Evaluation of a Novel PET Radioligand for Phosphodiesterase-4D (PDE4D)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 190064; 19-M-0064
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2020-02

CONDITIONS: Depression
Keywords: Healthy Control Subjects; PET Imaging; Receptor Occupancy; Depression
MeSH Terms: conditions — Depression | interventions — BPN14770

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Whole body PET Scan with intravenous 11C-T-1650 (Experimental): 10 mCi of 11C-T-1650 given intravenously once followed by a Whole Body PET scan. This was done for whole body dosimetry calculations.
  Interventions: Drug: [C-11]T-1650
- Brain PET scan with 11C-T-1650 and blocking with BPN14770 (Experimental): Baseline brain PET scan (scan 1) with 20 mCi of 11C-T-1650 given intravenously, followed by a second Brain PET scan (scan 2) 90-180 minutes after first dose administration of BPN14770 50mg given orally. A third brain PET scan (scan 3) is performed after the last dose of BPN14770. 20 mCi of 11C-T-1650 is given intravenously with each PET scan. BPN14770 50mg given orally twice a day for a total of seven doses. BPN14770 is a PDE4D-inhibitor.
  Interventions: Drug: [C-11]T-1650; Drug: BPN14770

INTERVENTIONS:
Drug: [C-11]T-1650 — radio-labeled drug
Drug: BPN14770 — selective compound
  Arms: Brain PET scan with 11C-T-1650 and blocking with BPN14770

SUMMARY:
Background:

The brain enzyme phosphodiesterase-4D (PDE4D) may affect thinking and depression. Drugs with some radioactivity can attach to enzymes and be seen on a scan. Researchers want to test a new radioactive drug, 11C-T-1650, to measure PDE4D in the brain and body. They also want to see if the new drug BPN14770 blocks 11C-T-1650 from the brain. They want to learn more about psychiatric disorders and possible treatments.

Objectives:

To study how well 11C-T-1650 helps show PDE4D on a scan and to see if BPN14770 blocks it.

Eligibility:

Healthy adults at least 18 years old

Design:

Participants will be screened in other protocols.

Some participants will have 1 body PET scan.

Some participants will have 2 brain PET scans and 1 brain MRI within 1 year.

Some participants (ages 18 55) will:

Have 3 brain PET scans and 1 MRI

Take BPN14770 by mouth twice daily for 3 7 days

Have blood and urine tests

Have a follow-up physical exam and heart test

PET (positron emission tomography) scans will take 2 3 hours. Participants will:

Have a thin plastic tube (catheter) placed in an arm vein by needle.

Get a small amount of 11C-T-1650 injected via catheter. Another catheter may be placed to draw blood.

Lie quietly on a bed that slides into a donut-shaped scanner without sleeping. They may get a short break.

Have heart and vital signs monitored.

Have blood and urine tests.

Learn about drinking fluids and urinating after the scan

MRI (magnetic resonance imagining) scans will take 30 60 minutes:

Participants will lie on a table that slides into a metal cylinder in a magnetic field.

Sponsoring Institute: National Institute of Mental Health

...

DETAILED DESCRIPTION:
Objective

Phosphodiesterase type 4 (PDE4) metabolizes 3 <=,5 <=-cyclic adenosine monophosphate (cAMP), thereby terminating this second messenger. PDE4 is selective to cAMP over cyclic guanosine monophosphate. PDE4 has four isozymes A, B, C, and D and basic studies suggest that type D (PDE4D) may play a key role in cognitive function and depression. That is, PDE4D inhibitors are expected to improve cognitive function and depressive symptoms.

In collaboration with Tetra Discovery Partners, we have developed a PET ligand, 11C-T-1650, to selectively image PDE4D. This type D selective ligand was developed based on 3D structural differences between PDE4D and PDE4 type B (PDE4B) Our PET studies using 11C-T-1650 in nonhuman primate have shown promising results, and we now seek to evaluate it in in healthy subjects.

This study has three primary objectives. First, we will determine whether the uptake of 11C-T-1650 in the brain reflects the distribution of PDE4D, as demonstrated by blocking with a PDE4D selective compound BPN14770, being developed by Tetra Discovery Partners for treating cognitive disorders including depression. Second, we will measure binding site occupancy of BPN14770 administered at doses that may be used in clinical trials. Third, we will measure the test/retest reproducibility of brain uptake quantified by kinetic modeling and using arterial blood samples.

Study Population

Healthy adult female and male volunteers (age greater than or equal to 18) will have either brain (n = 30) or whole body imaging (n = 10).

Design

* Phase 1: We will begin with whole body scanning in a single human subject using up to 10 mCi 11C-T-1650 The aim of this first scan will be to detect a tracer that disproportionately accumulates in a single radiosensitive organ, such as the gonads. If we confirm that radioactivity is fairly widely distributed in the body, higher activities may be injected.
* Phase 2: Fifteen healthy subjects will have three brain PET scans using 20 mCi of 11C-T-1650. Scan 1 will serve as the baseline scan for comparison to enzyme occupancy studies (Scan 2 and - Scans 2 and 3 will be enzyme occupancy studies using the PDE4D selective medication BPN14770.Scans 2 and Scan 3 will be performed approximately 90-180 min after the first dose of BPN14770 and after three-day administration, respectively. Scan 3 will be performed approximately 90-180 min after the last dose of the three-day administration of BPN14770. The dose of BPN14770 is 50 mg BID for three days, and a single dose on the fourth day. Comparison between Scan 1 and 2 provides accurate measurement of nonspecific binding of 11C-T-1650. Comparison between Scan 1 and 3 provides enzyme occupancy at a stable plasma concentration of BPN14770 based on Phase 1/2 clinical trials performed by Tetra Discovery Partners. Blood samples will be measured for BPN14770 levels.
* Phase 3: To obtain dosimetry information, we will perform a whole body PET scan using 11C-T-1650 (20 mCi) in up to nine healthy subjects.
* Phase 4: Fifteen healthy subjects will have two brain PET scans using 20 mCi of 11C-T-1650 to study test/retest reproducibility of the PET measurement. BPN14770 will not be administered in Phases 1, 3 or 4.

Outcome Measures

For whole body imaging, organ uptake will be quantified as a Standardized Uptake Value (SUV), which normalizes for injected activity and body weight. For Scan 1 and 2 of Phase 2 and all scans of Phase 4, uptake will be quantified as total distribution volume (VT) calculated with kinetic modeling and serial concentrations of parent radioligand in arterial plasma. For Scan 3 of Phase 3, brain uptake (SUV) normalized to plasma concentrations of 11C-T-1650 will be used to measure radioligand binding because the interval between Scan 2 and 3 is too short to repeat placing arterial line. From VT or normalized SUV, occupancy of BPN14770 and nonspecific binding of 11C-T-1650 will be measured. Occupancy of PDE4D will be compared to blood levels of BPN14770.

ELIGIBILITY:
* INCLUSION CRITERIA:

All phases

1. Age greater than equal 18.
2. Able to give written informed consent.
3. Medically and psychiatrically healthy.
4. Enrolled in 01-M-0254 The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers (PI: Dr. Carlos Zarate) or 17-M-0181 Recruitment and Characterization of Healthy Research Volunteers for NIMH Intramural Studies (PI: Dr. Joyce Chung).

Additional inclusion criterial for Phase 2

1. Age less than or equal to 55.
2. Body mass index between 18 kg/m2 to 32 kg/m2, inclusive, and body weight of greater than equal 50 kg (110 pounds).
3. Female subjects must be surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months prior to dosing of BPN14770), at least two years post-menopausal, or willing to use two barrier methods of contraception from initial screening until one month after taking the last dose of study drug.
4. Male subjects must be willing to inform female partners of their participation in the study and must agree to use adequate contraceptive methods (vasectomy performed at least 6 months prior to dosing BPN14770 or use at least one barrier method of birth control).

EXCLUSION CRITERIA:

All phases

1. Clinically significant laboratory abnormalities based on the following tests (performed under screening protocol 01-M-0254 or 17-M-0181): CBC; acute care panel; hepatic panel; mineral panel; urinalysis; urine drug screen; urine pregnancy test (females); and lipid panel; hepatitis panel (A, B, C); syphilis screening test; total protein; uric acid;creatine kinase; cholesterol; thyroid panel; prothrombin and partial prothrombin tests; and EKG.
2. Have a brain disease (such as multiple sclerosis or stroke).
3. Any current Axis I diagnosis, based on interview and self-reporting performed under screening protocol 01-M-0254 or 17-M-0181.
4. Positive HIV test.
5. Current or past history of significant cardiovascular, cerebrovascular, pulmonary, renal, or liver disease. Stable, well-controlled hypertension and hyperlipidemias are allowed.
6. Taking psychotropic drugs (i.e. benzodiazepines or antidepressants) including sedative antihistamines; moderate to strong inhibitors or inducers (i.e. fluconazole or ciprofloxacin) of any CYP450 enzyme. A complete listing of such inhibitors or inducers may be found in Attachment 1, List of P450 inhibitors.
7. Recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
8. Inability to lie flat on camera bed for at least two hours.
9. Pregnancy or breastfeeding.
10. Positive screen for drugs of abuse or cotinine (at screen or upon admission), or a positive alcohol result (upon admission).
11. Current use of psychiatric medications.
12. NIMH employees and staff or immediate family members of NIMH employee/staff.

Additional exclusion criterial for Phase 2 and 4

1. coagulation disorder;
2. thrombocytopenia;
3. Found to have inadequate collateral circulation of the radial artery
4. Are unable to have an MRI scan (e.g., pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments, metal fragments in the eye)

Additional exclusion criterial for Phase 2

1. Marked bradycardia (heart rate 45 beats per minute [bpm]) or tachycardia (heart rate 110 bpm) based on supine ECG values obtained at Screening, before the first dose of BPN14770 on the day of the study. Out-of-range vital signs may be repeated once at each eligibility assessment (prior to the start of dosing).
2. History of hematological disorders (e.g., thrombocytopenia) in the immediate family (i.e., parents and siblings).
3. Clinically important or significant conduction abnormalities on single ECG (including QTc interval 450 msec) or evidence or history of long QT syndrome. This exclusion applies to the ECGs obtained at Screening, before the first dose of BPN14770 on the day of the study.
4. Current or past history of gastric or duodenal ulcers or other diseases of the gastrointestinal tract that could interfere with absorption of study drug. Note: Subjects with a history of appendectomy or cholecystectomy may be enrolled.
5. Active acute or chronic infectious diseases.
6. Any history of alcohol or drug abuse within the previous year prior to the Screening visit (per the current edition of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition: DSM-5), or regular (daily) consumption of alcohol exceeding two bottles of beer, or the equivalent amount of other forms of alcohol (1 serving = 12 oz beer, 5.0 oz wine, or 1.5 oz distilled spirits).
7. Unwilling to abstain from alcohol within 72 hours of before the first dose of BPN14770.
8. Currently ingest nicotine in any way (including smoking cigarettes, vaping, and via patch), or have ingested any nicotine products within the past 3 months.
9. Participation in other clinical studies involving investigational drug within the previous 30 days prior to the first day of the study.
10. Unwilling to forgo donation of blood or blood products (including plasma) during the 8 weeks before the first day of the study.
11. History of allergy to penicillin or sulfonamides, or any other clinically significant drug allergy that includes symptoms such as shortness of breath, rash, or edema.
12. A suicidal ideation intensity score of 2 or higher per screening C-SSRS assessment and/or any suicidal behavior within the past 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-M-0064.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A single subject was enrolled only for pre-study whole body dosimetry calculations.
Period: Overall Study
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770 | Whole Body PET Scan With Intravenous 11C-T-1650
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770 | Whole Body PET Scan With Intravenous 11C-T-1650 | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Whole Brain Total Distribution Volume (VT) - Baseline
Description: To determine whether the uptake of 11C-T-1650 in brain reflects the distribution of PDE4D
Time Frame: 120 minutes after the start of the first scan
Population: The analyses included only those subjects who completed brain 11C-T-1650 and oral 50 mg BID of BPN14770 (twice/day, 7 times in total)
Measure: Mean (Standard Deviation); unit: mL x cm^3
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770
Number analyzed (Participants) | 2
mL x cm^3 | 8.2 (0.91)

2. Primary Outcome: Whole Brain Total Distribution Volume (VT)-1st Blocked
Description: To determine whether the uptake of 11C-T-1650 in brain reflects the distribution of PDE4D
Time Frame: 120 minutes after the start of the second scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL x cm^3
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770
Number analyzed (Participants) | 2
mL x cm^3 | 5.5 (20.2)

3. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (60-120min)-Baseline Whole Brain
Description: Measure binding site occupancy of BPN14770 administered at doses that may be used in clinical trials.
Time Frame: 120 minutes after the start of the scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770
Number analyzed (Participants) | 2
SUV x min | 102.1 (31.7)

4. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (60-120min)-1st Blocked Whole Brain
Description: Measure binding site occupancy of BPN14770 administered at doses that may be used in clinical trials.
Time Frame: 120 minutes after the start of the first scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770
Number analyzed (Participants) | 2
SUV x min | 71.719845 (20.2)

5. Primary Outcome: Standard UptakeValue (SUV) Area Under the Curve (AUC) (60-120min)-2nd Blocked Whole Brain
Description: Measure binding site occupancy of BPN14770 administered at doses that may be used in clinical trials.
Time Frame: 120 minutes after the start of the first scan
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SUV x min
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770
Number analyzed (Participants) | 2
SUV x min | 87.77384 (19.7)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770 | Whole Body PET Scan With Intravenous 11C-T-1650
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brain PET Scan With 11C-T-1650 and Blocking With BPN14770 (N=2) | Whole Body PET Scan With Intravenous 11C-T-1650 (N=1)
Polyuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03861000/Prot_SAP_000.pdf